CLINICAL TRIAL: NCT04930757
Title: Involvement of Polymorphonuclear Neutrophils and Platelets in Severe Form of COVID-19
Acronym: NeutroVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP210061
Record Dates: First submitted 2021-05-14; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Covid19; Neutrophils; Platelet aggregation activation; Clinical scores; SAPS II ("simplified acute physiology"); SOFA ("Sequential Organ Failure Assessment"); Global respiratory and non-respiratory scores
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with SARS-CoV-2 infection confirmed by RT-PCR from a nasopharyngeal swab.: Patients hospitalized in intensive care with SARS-CoV-2 infection confirmed by RT-PCR from a nasopharyngeal swab.

SUMMARY:
The main objective is to quantify the population of reverse migrating neutrophils in patients with COVID-19.

DETAILED DESCRIPTION:
This is a non-interventional transversal research whose main objective is to quantify the population of reverse migrating neutrophils in patients with COVID-19.

Design:

A multicentric (3 sites) clinical trial

Sample size :

200 patients

Population concerned:

Patients hospitalized in intensive care with SARS-CoV-2 infection confirmed by RT-PCR from a nasopharyngeal swab.

Duration of participation (treatment + follow-up): until the patient is discharged from the ICU and within 2 months top.

No interim analysis is planned. Analysis will be performed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care units of Saint-Antoine, Tenon and Pitié-Salpêtrière hospitals (Paris, France)
* With moderate to severe respiratory distress syndrome and SARS-CoV-2 infection confirmed by RT-PCR from a nasopharyngeal swab
* informed and not opposed to participation in research
* included within 4 hours following the paatient's admission

Exclusion Criteria:

* Patients under guardianship / curatorship
* Patients under AME

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in intensive care with SARS-CoV-2 infection confirmed by RT-PCR from a nasopharyngeal swab.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of circulating neutrophils in reverse migration | Within 4 hours following the patient admission in Intensive Care Units (ICU).
  Percentage of circulating neutrophils in reverse migration determined on a sample taken during the admission of COVID 19 patients to Intensive Care Units by flow cytometry: the samples will be incubated for 45 minutes with anti-human CXCR1, CD11c, CD11b, and CD62L antibodies. Erythrocytes will be lysed and fixed leukocytes will be analyzed by flow cytometry.

SECONDARY OUTCOMES:
Analysis of neutrophils and platelets | Within 4 hours following the patient admission in Intensive Care Units (ICU).
  The analysis of neutrophils and platelets, and of the inflammatory environment will be carried out on a sample taken on admission of patients to Intensive Care Units
  1. Phenotypic and functional analysis of neutrophils
     * Measurement of the oxidative explosion
     * Measurement of neutrophil apoptosis
     * Measurement of intravascular NETosis
  2. Analysis of platelet aggregation and activation
     * Quantification of the fraction of immature platelets (IPF)
     * Contribution of platelets to clot stiffness
     * ELISA assay of soluble platelet activation markers
     * Measurement of D-Dimers, von Willebrand factor, thrombin-antithrombin complex (TAT), α2-Plasmin-Plasmin-inhibitor
SAPS II score | From admission to the follow-up visits (Day 3, Day 7 and as part of usual care every 7 days until the patient is discharged and within 2 months top).
  Assessment of the link between phenotypic and functional markers of neutrophils on admission to the ICU.
  The severity of the disease is determined using clinical scores (SAPS II ("simplified acute physiology") and SOFA ("Sequential Organ Failure Assessment") (global SOFA, respiratory and non-respiratory) scores; these scores will be assessed during the period of hospitalization in Intensive Care Units. An association between these 2 scores (SAPSII and SOFA scores) and the neutrophil markers will be sought.
SOFA score | From admission to the follow-up visits (Day 3, Day 7 and as part of usual care every 7 days until the patient is discharged and within 2 months top).
  Assessment of the link between phenotypic and functional markers of neutrophils on admission to the ICU.
  The severity of the disease is determined using clinical scores (SAPS II ("simplified acute physiology") and SOFA ("Sequential Organ Failure Assessment") (global SOFA, respiratory and non-respiratory) scores; these scores will be assessed during the period of hospitalization in Intensive Care Units. An association between these 2 scores (SAPSII and SOFA scores) and the neutrophil markers will be sought.
Mortality rate | 2 months
  The mortality occurring within 2 months of admission of patients to an ICU will also be assessed.

OTHER OUTCOMES:
Quantification of the systemic inflammatory response upon admission to the ICU. | Within 4 hours following the patient admission in Intensive Care Units (ICU).
  Circulating levels of proinflammatory cytokines (IL-1bêta, IL-6, IL-8, TNFalpha, TGFbêta, IFNgamma, IL-17, IL-21, IL-22, IL-23, and IL-10) will be measured by Luminex and the levels of soluble adhesion molecules and in particular of soluble JAM-C and soluble mediators will be measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Hafid AIT-OUFELLA, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Intensive care department, Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided